CLINICAL TRIAL: NCT03008837
Title: Feasibility Study: fMRI Evaluation of Auricular PENFS for Fibromyalgia
Acronym: fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2113-M; 1IK1RX002113-01A2 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2017-01-04 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Percutaneous electrical neural field stimulator (PENFS) using the military field stimulator, a device that uses small needles inserted in the ear (like auricular acupuncture), which are connected by electrodes to a battery pack that is attached externally using adhesive to the back of the ear. The stimulator is meant to stimulate branches of the cranial nerves via the ear.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PENFS (Experimental): Veterans with fibromyalgia who meet study criteria and are randomized to the experimental group will receive standard therapy in addition to percutaneous electrical neural field stimulation (PENFS), which involves placement of small electrodes through a similar process to ear acupuncture to the ear. These electrodes are attached to a battery pack that is taped behind the ear and worn for 5-day intervals. The intention of this FDA-approved device is to relieve pain, though data on its effectiveness is still limited. Device placement (series of 4, weekly) will be performed by an Anesthesiology Pain Clinic provider. fMRI evaluation of neural changes, assessment of function and quality of life improvements will be performed at the beginning and end of the study.
  Interventions: Device: Military Field Stimulator
- Standard Therapy (Active Comparator): Veterans with fibromyalgia who meet study criteria and are randomized to standard therapy will receive physical therapy, medication management through the Anesthesiology Pain Clinic, and referral to a pain psychologist. fMRI evaluation of neural changes, assessment of function and quality of life improvements will be performed at the beginning and end of the study.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Device: Military Field Stimulator — The Military Field Stimulator (MFS/Neuro-Stim System), a percutaneous electrical neural field stimulation (PENFS) device evolved from PENS, is currently employed by the United States (US) military and used in the VA (contract number V797D-50453). There is some evidence based on a small trial of 20 postoperative patients that suggests PENS may have greater benefit than acupuncture for acute pain.
  Other Names: MFS, Neuro-Stim System, PENFS
  Arms: PENFS
Other: Standard Therapy — Standard therapy for fibromyalgia will include physical therapy, medication management through the Anesthesiology Pain Clinic, and referral to a pain psychologist.
  Arms: Standard Therapy

SUMMARY:
Given recent increasing opioid-related deaths and evidence showing against the use of opioids for non-malignant chronic pain, there is growing need for non-narcotic pain management. Fibromyalgia is a difficult to treat chronic pain condition that is often treated with opioids despite existing evidence. The prevalence of fibromyalgia is increased among Veterans returning from the gulf war and is already a significant burden in senior Veterans who may have suffered with chronic pain for decades already. Many treatment options for fibromyalgia carry intolerable side effects. PENFS (percutaneous electrical neural field stimulation) is a FDA-approved, non-pharmacologic therapy that is currently utilized within the military and VA system, but sufficient evidence regarding its outcomes and neural mechanisms have not been adequately investigated. An understanding of its neural underpinnings and analgesic effects could lead to 1) improvements in pain management and quality of life, 2) cost-savings and 3) development of new techniques to address pain.

DETAILED DESCRIPTION:
BACKGROUND: Fibromyalgia is a chronic pain syndrome that consists of chronic widespread pain, decreased physical function, fatigue, psychoemotional/sleep disturbances, and various somatic complaints, affecting anywhere from 5-10 million Americans, with ~1,500 Veterans carrying a diagnosis of fibromyalgia seen per year at the Atlanta VAMC alone. It is estimated that fibromyalgia costs the American population over $20 billion/year in lost wages and disability. Initial therapies often include complementary and alternative medicine (CAM) therapies, which are generally considered safe, although their efficacy has not been thoroughly evaluated for fibromyalgia. Thus, non-pharmacologic alternatives require more rigorous scientific investigation for the treatment of fibromyalgia. There is evidence to support the use of percutaneous electrical neural stimulation (PENS) in the treatment of pain conditions, which may have increased effects relative to acupuncture based on systematic reviews. While fMRI data for acupuncture and fibromyalgia exists, no such data exists for PENS treatment. An evolved form of PENS, percutaneous electrical neural field stimulation (PENFS) of the auricle is already used in the military and VA systems for the treatment of chronic pain, but evidence regarding its mechanisms and effects is lacking. Stimulation of the vagus nerve, which has auricular branches, has been previously studied for pain relief in fibromyalgia. However, application of PENS-type stimulation to the auricle has not been previously studied with fMRI, and this type of therapy may lead to neural changes worthy of further exploration. OBJECTIVE: To evaluate the feasibility of using fMRI as a biomarker for the neural substrates of pain and functional changes following PENFS treatments. HYPOTHESIS: PENFS will result in decreased functional connectivity between the insula and default mode network as evaluated by fMRI, which will correlate to more significant improvements in pain and function relative to standard therapy for fibromyalgia. METHODS: Subjects who meet study criteria will receive baseline assessments including resting state fMRI, collection of biobehavioural information such as cognitive and psychological assessments on standardized forms, eating, sleeping and drinking habits, Defense and Veterans Pain Rating Scale (DVPRS), arm curl, 30-s chair stand, and pain interference scores. Subjects will be stratified based on age and gender and then divided into standard therapy control (medication management and physical therapy) or PENFS (series of 4, weekly) treatments and assessed for fMRI changes 2 weeks after the final treatment. Pain and function will also be assessed at the 2 weeks, 6 weeks and 12 weeks following the final treatment. CLINICAL RELEVANCE: Auricular PENFS has not been studied with fMRI. Stimulation of the auricle may produce neural changes that differ from traditional therapies. Understanding the underlying neural mechanisms of auricular PENFS could assist in developing targeted treatments for fibromyalgia and chronic pain. Further, if PENFS can significantly improve pain relief and function over standard therapies, it could decrease the need for opioid analgesics and their associated risks, which is a primary objective of the VA Opioid Safety Initiative. The present investigation will not only serve to elucidate neural changes with PENFS, but could be directly applicable to our Veterans suffering from fibromyalgia by providing evidence regarding the relative effectiveness of this already clinically-employed non-pharmacologic treatment (or lack thereof), and result in evidence-based implementation and potential cost savings to the VA system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male and female Veterans age 20-60 with a diagnosis of fibromyalgia as diagnosed by a clinician, by chart review, and by the most recent American College of Rheumatology 2010 criteria for the diagnosis of fibromyalgia. 70,71
* Subjects must self-report consistent, daily pain (greater than 5 on the VAS) >90 days.
* Subjects must have intact skin free of infection at the site of implantation.
* Subjects must be willing to participate and understand the consent.
* Subjects must be right-handed in order to provide consistency in brain structure and function.

Exclusion Criteria:

* Subjects must not be currently pregnant, since effects of fMRI and electrical current on the developing fetus are not well-known.
* Subjects must not have an implanted electrical device such as a vagal stimulator, pacemaker, or spinal pain pump, which are not compatible with MRI.
* Subjects must not have a history of seizures or neurologic condition that may alter the structure of the brain.
* Subjects must not have a history of drug abuse or severe, uncontrolled psychiatric illness such as schizophrenia or major depressive disorder with suicidal ideation.
* Subjects must not have psoriasis vulgaris or other skin conditions that may increase the risk of infection at the implantation site.
* Subjects must not have severe anxiety, claustrophobia, or other conditions that may prevent their ability to lie at rest in an MRI scanner. This will be determined after discussion with the patient regarding their own perceived ability to lie at rest in an MRI scanner without the use of additional sedating medications.
* Subjects must not introduce new medications or treatments for fibromyalgia symptoms during the course of the study to prevent confounding results.
* Subjects must not have a concurrent autoimmune or inflammatory disease that causes pain such as systemic lupus erythematosus, inflammatory bowel disease or rheumatoid arthritis, since this could decrease the effect of treatment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Woodbury, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gebre M, Woodbury A, Napadow V, Krishnamurthy V, Krishnamurthy LC, Sniecinski R, Crosson B. Functional Magnetic Resonance Imaging Evaluation of Auricular Percutaneous Electrical Neural Field Stimulation for Fibromyalgia: Protocol for a Feasibility Study. JMIR Res Protoc. 2018 Feb 6;7(2):e39. doi: 10.2196/resprot.8692. PMID 29410385
- [Derived] Woodbury A, Krishnamurthy V, Gebre M, Napadow V, Bicknese C, Liu M, Lukemire J, Kalangara J, Cui X, Guo Y, Sniecinski R, Crosson B. Feasibility of Auricular Field Stimulation in Fibromyalgia: Evaluation by Functional Magnetic Resonance Imaging, Randomized Trial. Pain Med. 2021 Mar 18;22(3):715-726. doi: 10.1093/pm/pnaa317. PMID 33164085
- See also: Peri-Auricular PENFS for Chronic Pain — http://article.sapub.org/10.5923.j.cmd.20150504.03.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 veterans were initially consented. However, 6 of these veterans either could not begin the study within the study period, moved out of state, or received implanted MRI-incompatible devices that excluded them from the study following the initial consent, but prior to randomization.
Groups:
- PENFS: Veterans with fibromyalgia who meet study criteria and are randomized to the experimental group will receive standard therapy in addition to percutaneous electrical neural field stimulation (PENFS), which involves placement of small electrodes through a similar process to ear acupuncture to the ear. These electrodes are attached to a battery pack that is taped behind the ear and worn for 5-day intervals. The intention of this FDA-approved device is to relieve pain, though data on its effectiveness is still limited. Device placement (series of 4, weekly) will be performed by an Anesthesiology Pain Clinic provider. fMRI evaluation of neural changes, assessment of function and quality of life improvements will be performed at the beginning and end of the study.
  Military Field Stimulator: The Military Field Stimulator (MFS/Neuro-Stim System), a percutaneous electrical neural field stimulation (PENFS) device evolved from PENS, is currently employed by the United States (US) military
Period: Overall Study
Arm/Group | PENFS | Standard Therapy
Started | 12 | 9
Completed | 9 | 5
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PENFS | Standard Therapy | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Full Range); unit: years] | 50 [33 to 60] | 48.56 [32 to 60] | 49.35 [32 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 9 | 21
DVPRS (Pain) [Mean (Standard Deviation); unit: units on a scale] — pain measure that includes a 0-10 scale where 0 means no pain and 10 means greatest pain imaginable
  units on a scale | 6.42 (0.84) | 8 (0.77) | 7.41 (1.35)

OUTCOME MEASURES:

1. Primary Outcome: fcMRI as a Biomarker to Investigate Functionally Correlated Neural Substrates of Pain in Patients Undergoing PENFS
Description: 2 weeks following the final treatment, subjects in the PENFS group were be evaluated for changes in functional connectivity between the right posterior insula seed and other areas of the DMN as evaluated by fcMRI relative to standard treatment controls, using whole brain analysis. The measurement is increase/decrease of signal in a given region, thresholded at p <0.05, summarized into a value representing 'size of region of increase' or 'size of region of decrease' after subjects scans were combined/mapped onto a standard MNI brain. Only clusters of over 40 voxels were included, and the size of the region is reported in voxel size. The averaged brains for baseline fcMRI was subtracted from post-treatment for each group, and then these averaged differences were subtracted from each other. While other areas of the brain met threshold criteria in the analysis, only areas belonging to the DMN are reported.
Time Frame: baseline and 2 weeks post-treatment
Population: Using a right posterior insula seed for seed-based whole-brain analysis in AFNI, a difference of the differences was measured. Clusters greater than 40 voxels in size with p<0.05 (set in AFNI) found in the default mode network (DMN) are included in the outcome table.
Measure: Number; unit: Cluster size (voxels)
Groups:
- PENFS (Post-pre): Veterans with fibromyalgia who meet study criteria and are randomized to the experimental group will receive standard therapy in addition to percutaneous electrical neural field stimulation (PENFS). This column shows the number of voxels in clusters that showed increased or decreased connectivity following treatment, >40 voxel clusters, thresholded at p<0.05 in AFNI.
- Standard Therapy Control (Post-pre): Veterans with fibromyalgia who meet study criteria and are randomized to the control group will receive standard therapy including medications and physical therapy. This column shows the number of voxels in clusters that showed increased or decreased connectivity following standard therapy, >40 voxel clusters, thresholded at p<0.05 in AFNI.
Arm/Group | PENFS (Post-pre) | Standard Therapy Control (Post-pre)
Number analyzed (Participants) | 9 | 7
Cluster size (voxels)
  Anterior cingulate (L) | 0 | 0
  Inferior parietal lobule (R) | 0 | 0
  Posterior cingulate cortex (L) | 0 | 61
Statistical Analysis 1: Comparison: PENFS (Post-pre) vs Standard Therapy Control (Post-pre); PENFS (post-pre) - Standard Therapy (post-pre); Test type: Other — Using seed-based analysis with a right posterior insula seed, cluster size was set at 40 voxels, and p-value was thresholded at p<0.05 to compare the differences between the two groups in terms of connectivity between the right posterior insula and areas of the DMN identified based on a priori hypotheses; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 40 — Standard therapy control (post-pre) was subtracted from PENFS (post-pre)

2. Secondary Outcome: Change in Defense Veterans Pain Rating Scale (DVPRS) From Baseline
Description: For fibromyalgia patients, pain will be assessed in the PENFS group relative to standard treatment controls, as indicated by analgesic Defense and Veterans Pain Rating Scale (DVPRS) at 2, 6 and 12 weeks follow-up. This is a validated pain measure that includes a 0-10 scale where 0 means no pain and 10 means greatest pain imaginable. Higher scores indicate worse reported pain outcomes.
Time Frame: 2, 6 and 12 weeks follow-up
Population: Not all individuals presented for all follow-up visits, but all participants included in the analysis were present for baseline assessments, pre- and post- imaging studies, and at least one follow-up visit. Missing data was not imputed and not used for analysis in order to avoid distortions related to imputation in the small sample size.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PENFS | Standard Therapy
Number analyzed (Participants) | 9 | 7
score on a scale
  2 weeks | -0.9 [-4.4 to 2.6] | -1.4 [-8.8 to 6]
  6 weeks: number analyzed (Participants) | 8 | 6
  6 weeks | -1.1 [-5.1 to 2.9] | -0.5 [-2.6 to 1.6]
  12 weeks: number analyzed (Participants) | 9 | 5
  12 weeks | -1.3 [-5.3 to 2.7] | -0.1 [-3.4 to 3.2]

3. Secondary Outcome: Change in Pain Interference With "Activity," "Sleep," "Mood", and "Stress" From Baseline
Description: Pain interference scores were measured using supplemental questions on the Defense and Veterans Pain Rating Scale (DVPRS). Participants were asked to evaluate on a scale of 0-10 the level to which pain interfered with their "activity," "sleep," "mood", and "stress," with 10 being the worst interference, and 0 being no interference.
Time Frame: 2, 6 and 12 weeks follow-up
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PENFS | Standard Therapy
Number analyzed (Participants) | 9 | 7
score on a scale
  2 weeks - Activity | -1.2 [-4.7 to 2.3] | 0.9 [-8 to 9.8]
  2 weeks - Sleep | -1.6 [-7.4 to 4.2] | -0.4 [-11.7 to 10.9]
  2 weeks - Mood | -1 [-6.1 to 4.1] | -0.6 [-11.1 to 9.9]
  2 weeks - Stress | -1.4 [-5 to 2.2] | 0 [-9.7 to 9.7]
  6 weeks - Activity: number analyzed (Participants) | 8 | 6
  6 weeks - Activity | -1.2 [-5.7 to 3.3] | 1.2 [-1.9 to 4.3]
  6 weeks - Sleep: number analyzed (Participants) | 8 | 6
  6 weeks - Sleep | -1.6 [-7.1 to 3.9] | 1.8 [-2.4 to 6]
  6 weeks - Mood: number analyzed (Participants) | 8 | 6
  6 weeks - Mood | -1.4 [-6.7 to 3.9] | 1.8 [-2.7 to 6.3]
  6 weeks - Stress: number analyzed (Participants) | 8 | 6
  6 weeks - Stress | -1.8 [-6.2 to 2.6] | 1.7 [-1.9 to 5.3]
  12 weeks - Activity: number analyzed (Participants) | 9 | 5
  12 weeks - Activity | -1.6 [-6.3 to 3.1] | 1 [-6.2 to 8.2]
  12 weeks - Sleep: number analyzed (Participants) | 9 | 5
  12 weeks - Sleep | -1.7 [-6.3 to 2.9] | 2.2 [-3.7 to 8.1]
  12 weeks - Mood: number analyzed (Participants) | 9 | 5
  12 weeks - Mood | -2.1 [-6.4 to 2.2] | 1.8 [-5.5 to 9.1]
  12 weeks - Stress: number analyzed (Participants) | 9 | 5
  12 weeks - Stress | -1.9 [-5.2 to 1.4] | 1.8 [-4.6 to 8.2]

4. Secondary Outcome: Change in Number of Bicep Curls From Baseline (Left Arm)
Description: Objective tests for functional improvement will be performed at 2, 6, and 12 weeks follow-up and include 30 sec chair stand tests. The total number of full bicep curls (left arm) participants could perform using were measured over a 30-second period at each visit.
Time Frame: 2, 6 and 12 weeks follow-up
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: bicep curls
Arm/Group | PENFS | Standard Therapy
Number analyzed (Participants) | 9 | 7
bicep curls
  2 weeks | 4.6 [-8.1 to 17.3] | 1.7 [-12 to 15.4]
  6 weeks: number analyzed (Participants) | 8 | 6
  6 weeks | 6.1 [-7 to 19.2] | -1.8 [-14.2 to 10.6]
  12 weeks: number analyzed (Participants) | 9 | 5
  12 weeks | 5.8 [-7.4 to 19] | 0 [-15.5 to 15.5]

5. Secondary Outcome: Change in Number of Bicep Curls From Baseline (Right Arm)
Description: Objective tests for functional improvement will be performed at 2, 6, and 12 weeks follow-up and include 30 sec chair stand tests. The total number of full bicep curls (right arm) participants could perform using were measured over a 30-second period at each visit.
Time Frame: 2, 6 and 12 weeks follow-up
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: bicep curls
Arm/Group | PENFS | Standard Therapy
Number analyzed (Participants) | 9 | 7
bicep curls
  2 weeks | 4.2 [-5.8 to 14.2] | 0.7 [-14.4 to 15.8]
  6 weeks: number analyzed (Participants) | 8 | 6
  6 weeks | 6 [-8.4 to 20.4] | 0.8 [-12.4 to 14]
  12 weeks: number analyzed (Participants) | 9 | 5
  12 weeks | 4.6 [-8.7 to 17.9] | 0.2 [-11.2 to 11.6]

6. Secondary Outcome: Change in Sit-to Stand Test From Baseline
Description: Objective tests for functional improvement will be performed at 2, 6, and 12 weeks follow-up and include 30 sec chair stand tests. The total number of full sit-to-stands participants could perform were measured over a 30-second period at each visit.
Time Frame: 2, 6 and 12 weeks follow-up
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: sit-to-stands
Arm/Group | PENFS | Standard Therapy
Number analyzed (Participants) | 9 | 7
sit-to-stands
  2 weeks | 2.7 [-3.9 to 9.3] | 0.3 [-7.8 to 8.4]
  6 weeks: number analyzed (Participants) | 8 | 6
  6 weeks | 3.1 [-6.6 to 12.8] | 0.3 [-7.8 to 8.4]
  12 weeks: number analyzed (Participants) | 9 | 5
  12 weeks | 1.7 [-7 to 10.4] | 1.4 [-6.3 to 9.1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PENFS | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 2/12 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PENFS (N=12) | Standard Therapy (N=9)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0 — Minor skin irritation reported at implantation site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03008837/Prot_SAP_000.pdf